CLINICAL TRIAL: NCT03893604
Title: Comparing the Effects of tDCS on Endurance Parameters Between High Level and Recreational Athletes
Brief Title: Effects of tDCS on High Level and Recreational Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2017-313
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Athlete
Keywords: tDCS; Athlete; Isokinetic; Endurance; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, sham-controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The device is preprogrammed by a third party non participating in any element in the study. They then chose (using opaque envelopes) the treatment code for each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): Subjects will receive 20min anodal tDCS
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of Sham anodal tDCS
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 20 minutes of anodal tDCS (C3/FP2) 2mA or sham
  Other Names: Non invasive brain stimulation

SUMMARY:
Healthy recreational and high level athletes will undergo 2 randomized, cross-over counterbalanced sessions of anodal tDCS or sham tDCS.

The primary outcome is an isokinetic evaluation of their hamstrings' and quadriceps' endurance after each session

DETAILED DESCRIPTION:
Recruitment :

Healthy recreational and high level athletes will be recruited through social media and advertisements.

Each subject came twice to the Liege University Hospitals' isokinetic lab. Each session began with strapping the subjet into the isokinetic machine, making sure that all the settings were adapted to the subject. Then, each subject received either anodal tDCS, of sham tDCS. Neither the evaluator or the subject knew which they were receiving. Immediately following tDCS, there was a warmup consisting of stationary bike, and an isokinetic warmup. Then, subjects' endurance was using a maximal isokinetic tests, at 30 maximal concentric and eccentric contractions at a speed of 180°/s.

ELIGIBILITY:
Inclusion Criteria:

* For the "recreational" group at most 3 hours of sport a week
* For the "athletic" group, at least 10 hours of sport a week
* Right handed and footed

Exclusion Criteria:

* One on the TSST (in high and relatively high risk sections)
* Previous neurological or orthopedic pathologies affecting limbs

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Peak Strength | Immediately after tDCS and sham
  Peak strength (measured by the isokinetic machine) is measured after each of the 30 repetitions.
  Peak strength of the 30 repetitions will be measured, and how strength decreases throughout the test will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bornheim, Msc, Principal Investigator — Liege University Hospital
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No